CLINICAL TRIAL: NCT00498030
Title: Predicting Insulin Resistance in American Indian Youth
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: Indian Health Service (IHS) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 0453-04-FB; U26IHS300002/01 (Other Grant/Funding Number: Aberdeen Area Tribal Chairman's Health Board)
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Insulin Resistance; Stress, Psychological
Keywords: Insulin Resistance; Stress, Psychological
MeSH Terms: conditions — Insulin Resistance; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples are only retained until specific tests are completed. Some tests are done in the clinical lab and some tests are done in the research lab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify risks that may contribute to increased insulin resistance which may help explain some of the increased incidence of type 2 diabetes in American Indian Youth, at the Rosebud reservation ages 5 to 18 years old. If specific positive indicators of insulin resistance are present, individuals are recruited back in one year for repeat of all measures.

DETAILED DESCRIPTION:
Type 2 diabetes is rapidly becoming more prevalent in the United States but especially among minority populations at a younger age. Identification of risk factors, including traditional risk factors such as increased BMI, lack of exercise, increased glucose in the diet, higher blood pressure and lipids, along with other factors such as chronic stress, use of alcohol or other drugs has not previously been done with minority youth. If risk factors can be identified, more strategies for prevention of diabetes can be developed that specifically target this population. This study will enroll 300 Native American Youth over a 4 year period and perform body measurements including height, weight, waist circumference, blood pressure and lab values including a 2hour glucose tolerance test, fasting lipids, and a urine albumin creatinine ratio test. In addition, subjects will be asked to identify behavior and feelings of stress in everyday lives. Subjects who are determined to be at increased risk of developing diabetes will be asked to repeat the tests in one year. The results will be reported to the tribal council to help determine prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Native American youth between ages of 5 and 18 who are eligible for health care at Rosebud Sioux Reservation (Rosebud, SD) and willing to be measured and participate in a 2 hour glucose tolerance test and who have parental consent.

Exclusion Criteria:

* Those who have diabetes previously identified or those with chronic steroid use, or identified conditions that affect weight balance such as cancer.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Native American youth between ages of 5 and 18 who are eligible for health care at Rosebud Sioux Reservation (Rosebud, SD) and willing to be measured and participate in a 2 hour glucose tolerance test and who have parental consent.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2005-12-05 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Resistance | one year
  This study will assess for change in insulin resistance in Native American Children over one year.

SECONDARY OUTCOMES:
Changes in Body Mass Index (BMI) | One year
  To determine if BMI is a good marker for insulin resistance and if BMI changes after enrollment in diabetes intervention program.
Change in Fasting Lipids | One year
  To determine if fasting lipids levels are a good marker for insulin resistance and if fasting lipid levels change after enrollment in diabetes intervention program.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Larsen, MD, Principal Investigator — University of Nebraska
Locations (1):
- Rosebud Indian Reservation, Rosebud, South Dakota, United States

REFERENCES:
- [Result] Nsiah-Kumi PA, Beals J, Lasley S, Whiting M, Brushbreaker C, Erickson J, Qiu F, Yu F, Canaris G, Larsen JL. Body mass index percentile more sensitive than acanthosis nigricans for screening Native American children for diabetes risk. J Natl Med Assoc. 2010 Oct;102(10):944-9. doi: 10.1016/s0027-9684(15)30714-8. PMID 21053710
- [Result] Nsiah-Kumi PA, Lasley S, Whiting M, Brushbreaker C, Erickson JM, Qiu F, Yu F, Larsen JL. Diabetes, pre-diabetes and insulin resistance screening in Native American children and youth. Int J Obes (Lond). 2013 Apr;37(4):540-5. doi: 10.1038/ijo.2012.199. Epub 2012 Dec 11. PMID 23229738
- [Result] Nsiah-Kumi PA, Erickson JM, Beals JL, Ogle EA, Whiting M, Brushbreaker C, Borgeson CD, Qiu F, Yu F, Larsen JL. Vitamin D insufficiency is associated with diabetes risk in Native American children. Clin Pediatr (Phila). 2012 Feb;51(2):146-53. doi: 10.1177/0009922811417290. Epub 2011 Oct 20. PMID 22019791